CLINICAL TRIAL: NCT00403663
Title: Effect of Body Mass Index on the ED95 of Intrathecal Hyperbaric Bupivacaine for Elective Cesarean Section
Brief Title: Effect of Body Mass Index on the Dose of Intrathecal Hyperbaric Bupivacaine for Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-02; 06-0206-E
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pain; Obesity
Keywords: Body mass index; Combined Spinal-Epidural Anesthesia; Cesarean section; Obesity
MeSH Terms: conditions — Pain; Obesity | interventions — Bupivacaine; Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bupivacaine 0.75% with fentanyl and morphine — the following administered once, by spinal injection; 9-12 mg 0.75% hyperbaric bupivacaine 10 mcg fentanyl 100 mcg morphine

SUMMARY:
Combined spinal - epidural (CSE) anesthesia is a well established technique used for elective Cesarean section. As its name suggests, it combines two anesthesia techniques - spinal and epidural. Adjusting the dose of freezing medication for body size is not as simple as giving a larger dose to a larger person. This study asks a simple, yet important question: does your body mass index (BMI) influence the amount of freezing medication needed for adequate CSE anesthesia for Cesarean section? BMI is a number calculated from your height and weight. In patients with a higher BMI, freezing medication appears to spread farther (to a higher level) in the spinal fluid. When freezing is too high, it can cause unwanted side effects. Therefore, in order to provide optimal spinal anesthesia to patients with a higher BMI, it may be advisable to administer less freezing medication. In this study, we want to find the ideal dose of freezing medication for patients with a higher body mass index, and compare it to the dose found to be ideal for patients with normal body mass index.

DETAILED DESCRIPTION:
Spinal anesthesia is the most common anesthetic technique used for Cesarean section. It offers many advantages over epidural and general anesthesia. However, one of the limitations of spinal anesthesia in Obstetrics is the use of a single shot technique as the continuous technique is associated with unacceptable incidence of PDPH. It is difficult to predict the exact level of sensory block because many factors affect the spread of local anesthetic injected into the CSF. Theoretically, obese patients may have greater intra-abdominal pressure, leading to compression of the inferior vena cava and engorgement of the epidural venous plexus, which in turn increases the pressure inside the epidural space. This augmented pressure is transmitted to the dural sac and diverge the CSF from the lumbosacral region, leading to a decrease in CSF volume. It has been demonstrated that the volume of CSF in lumbosacral region is an important factor affecting intrathecal spread of anesthetics.

Our hypothesis is that obese women require less intrathecal hyperbaric bupivacaine than do normal weight women to achieve satisfactory surgical anesthesia for elective Cesarean section.Two groups of patients will be studied separately. Patients with BMI greater than or equal to 30 will be included in the obese group, also denominated study group. Patients with BMI less than 25 will be included in the normal weight group, also denominated control group. BMI will be calculated based on the patient's pre-pregnancy weight. For each group, the up-down sequential allocation method based on the Narayana rule will be used to find the minimum effective dose of intrathecal hyperbaric bupivacaine 0.75% associated with opioids necessary for satisfactory outcome in 95% of the pregnant women undergoing cesarean section, i.e. ED95.

There are two possible outcomes in our study: a satisfactory outcome is defined if the sensory block reaches at least at T6 and the patient does not complain of any pain or discomfort that requires intraoperative supplemental drugs; an unsatisfactory outcome is defined if the sensory block reaches a level lower than T6 or the patient complains of pain or discomfort that requires intraoperative supplemental drugs. The decision whether or not the supplementation is required will be made exclusively by the patient, and not by the physician in charge.

ELIGIBILITY:
Inclusion Criteria:

* Obese group: All pregnant women at term (over 37 weeks) scheduled for elective Cesarean section, with pre-pregnancy BMI greater than 30
* Normal weight group: All pregnant women at term (over 37 weeks) scheduled for elective Cesarean section, with pre-pregnancy BMI less than 25.

Exclusion Criteria:

* Patient's refusal.
* Patients with any absolute or relative contraindication for spinal/epidural anesthesia.
* Patients with BMI between 25 and 30.
* Patients with more than one fetus.
* Patients unable to communicate in English effectively.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the success/failure of the block. Success meaning a sensory block level at least at T6 within 15 minutes after intrathecal injection and no requirement of any supplemental analgesic by the patient throughout the CS. | 15 minutes

SECONDARY OUTCOMES:
Upper level of sensory blockage determined by the pinprick at midaxillary line | 60 minutes
VAPS during surgery | 60 minutes
Dose of lidocaine 2% required as supplementation | 60 minutes
Dose of IV fentanyl or ketamine required as supplementation | 60 minutes
Conversion to general anesthesia | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — Department of Anesthesia and Pain Management, Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada